CLINICAL TRIAL: NCT00592345
Title: High-Dose Proton/Photon RT + Surgery of Sarcomas of the Thoracic, Lumbar Spine/Sacrum
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tom DeLaney, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-502
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Mesenchymal Tumor
Keywords: sarcoma of the thoracic/lumbar/spine/sacrum; paraspinal soft tissues; proton radiation therapy; photon radiation therapy; radiation applicator plaque
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Proton Beam Radiation — Administered over a period of 12 weeks.
Radiation: Photon Beam Radiation — Administered over a period of 12 weeks.
Radiation: Interoperative radiation — Radioactive plaque applied at the time of surgical removal of the tumor.

SUMMARY:
The purpose of this study is to test the effectiveness of high dose radiation administered by both proton and photon therapy. Radiation is an effective treatment for many types of tumors and it is thought that radiation alone, when given in much higher doses over a shorter period of time, may be more effective in controlling recurrence of sarcoma.

DETAILED DESCRIPTION:
* In this study three types of radiation will be used: standard radiation (called photon); alternative form of radiation called proton beam therapy; and a localized radiation applicator plaque that can be applied to the surface of the dura (the fibrous outer envelope that surrounds the spinal cord and fluid surrounding the spinal cord) at time of surgical removal of the tumor.
* Radiation treatments (photon and proton) and possibly surgical removal of portions of the tumor with intraoperative radiation delivery to the surface dura with intraoperative radiation delivery will be performed over a period of 12 weeks. As part of the treatment planning process, participants will need two treatment planning CT scans and 2-3 treatment planning sessions.
* Participants will receive, in total, 39-43 photon/proton treatments.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of malignant mesenchymal tumor of the thoracic/lumbar/spine/sacrum or paraspinal soft tissues involving nerve roots or extending into spinal canal. Inter-osseous bone sarcomas are to be managed by wide resectional surgery for patients that are medically operable.
* Patient tumor status: 1) post biopsy or post resection with gross residual disease 2) post grossly complete resection but with margins positive or very close or tumor spill or cut through
* Lesion may be primary or recurrent after prior surgery
* No clinical, radiographic or other evidence of distant metastasis
* Fit for the exposure of the affected vertebral segment
* Life expectancy of greater than 36 months
* KPS equal to or greater than 70
* 18 years of age or older
* Declines radical surgery
* No prior radiation treatment to the affected spine region

Exclusion Criteria:

* Pregnancy
* Disease/conditions characterized by high radiation sensitivity. These include genetic diseases, such as ataxia telangiectasia. Major local conditions which are the local tolerance viz., multiple surgical procedures, serious local injuries.
* No evident cord/cauda malfunction for causes other than effects of local tumor growth or due to metabolic effects of tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1999-05; Primary Completion 2005-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To define the efficacy of high dose fractionated radiation alone or combined with surgery in this patient population. | 3 years

SECONDARY OUTCOMES:
To evaluate the acute and later tolerance in 50 patients of high dose proton/photon radiation treatment. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. DeLaney, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States